CLINICAL TRIAL: NCT01261806
Title: Mental Health Services for Toddlers in Foster Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Mary Dozier, UNIDEL-Amy E dupont Professor, Psychology, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NIH R01 MH052135
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Behavior Problems
MeSH Terms: conditions — Mental Disorders | interventions — butyl phosphorotrithioate; Occupational Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attachment and Biobehavioral Catch-up (Experimental): Attachment and Biobehavioral Catch-up: 10 session intervention in foster families' homes designed to enhance parental nurturance, synchrony, and provide skills such that parents can help children calm down when overwhelmed.
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up
- Developmental Education for Families (Active Comparator): 10 session intervention in foster families' homes that targets cognitive and motor skills of children
  Interventions: Behavioral: Developmental Education for Families

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up — Enhances nurturance, following the lead, and calming behaviors
  Other Names: ABC; ABC-T; Attachment and Biobehavioral Catch-up for Foster Toddlers
  Arms: Attachment and Biobehavioral Catch-up
Behavioral: Developmental Education for Families — Attention control: Enhances parents understanding of developmental milestones
  Other Names: DEF; Occupational Therapy/Physical Therapy
  Arms: Developmental Education for Families

SUMMARY:
Toddlers (2- to 3-year-old children) in foster care often have difficulty regulating behavior and biology, and are at risk for a host of mental health problems. Critical issues for toddlers straddle the challenges of infancy and preschool years. In particular, toddlers in foster care face significant challenges in forming new attachment relationships and developing behavioral and biological regulatory capabilities. This project will assess the effectiveness of an intervention that targets these issues. Attachment and Biobehavioral Catch-up for Toddlers in Foster Care (ABC-T) was developed to help parents: provide nurturing care so that children develop secure, trusting relationships; and supporting children when they become overwhelmed that enhance children's ability to regulate behavior and biology. This intervention's effectiveness will be assessed in a randomized clinical trial.

DETAILED DESCRIPTION:
This study assesses the efficacy of a 10-session intervention for young children in the foster care system. Children are randomly assigned to the experimental condition (ABC-T) or to a treatment control (DEF). In the Attachment and Biobehavioral Catch-up for Toddlers (ABC-T) condition, children's foster parents receive an intervention that focuses on nurturance, following children's lead, and helping children settle when they become overwhelmed. In the Developmental Education for Families (DEF) intervention, children's foster parents receive an intervention that focuses on enhancing children's cognitive and motor skills. Both of the interventions are provided in families' homes for 10 sessions of about 60 minutes duration. Outcomes include attachment (assessed in the Preschool Strange Situation), cortisol production (assessed diurnally), child behavior problems (assessed through laboratory procedures that stress children), and through psychiatric interviews.

ELIGIBILITY:
Inclusion Criteria:

* 2 -3 years of age, in foster care

Exclusion Criteria:

* Not in foster care

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2010-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Problem behaviors | Annual
  Assessed through laboratory measures of child behavior problems. (Disruptive Behavior Diagnostic Observation Schedule)

SECONDARY OUTCOMES:
Attachment | Once at post-intervention
  Assessed through Preschool Strange Situation

OTHER OUTCOMES:
Cortisol production | Annual
  Diurnal cortisol assessed through saliva sampling at wake-up and bedtime

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dozier, Ph.D., Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raby KL, Freedman E, Yarger HA, Lind T, Dozier M. Enhancing the language development of toddlers in foster care by promoting foster parents' sensitivity: Results from a randomized controlled trial. Dev Sci. 2019 Mar;22(2):e12753. doi: 10.1111/desc.12753. Epub 2018 Oct 3. PMID 30230658